CLINICAL TRIAL: NCT00003859
Title: Trial of Chemotherapy Utilizing Carboplatin, Vincristine, Cyclophosphamide and Etoposide for the Treatment of Central Nervous System Primitive Neurectodermal Tumors of Childhood
Brief Title: Surgery Plus Radiation Therapy With or Without Chemotherapy in Treating Children With Primitive Neuroectodermal Tumors of the CNS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Societe Internationale d'Oncologie Pediatrique (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067022; SIOP-PNET-III; EU-99003; UKCCSG-9102
Record Dates: First submitted 1999-11-01; First posted 2004-06-09 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2009-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood supratentorial primitive neuroectodermal tumor; recurrent childhood supratentorial primitive neuroectodermal tumor
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Carboplatin; Cyclophosphamide; Etoposide; Vincristine; Surgical Procedures, Operative; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: cyclophosphamide
Drug: etoposide
Drug: vincristine sulfate
Procedure: surgical procedure
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. It is not yet known whether undergoing surgery plus radiation therapy is more effective with or without chemotherapy for primitive neuroectodermal tumors of the CNS.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery plus radiation therapy with or without chemotherapy in treating patients who have primitive neuroectodermal tumors of the CNS.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine whether chemotherapy utilizing carboplatin, vincristine, cyclophosphamide, and etoposide improves the prognosis for children with primitive neuroectodermal tumors of the central nervous system when given after surgery and before radiotherapy. II. Assess prospective factors that may determine ultimate prognosis in this patient population. III. Determine the quality of survival of these patients on both treatment regimens.

OUTLINE: This is a randomized study. Patients undergo surgical removal of the primary tumor. Following surgery, patients are randomized to receive radiotherapy alone (arm I) or chemotherapy followed by radiotherapy (arm II). Arm I: Patients begin receiving radiotherapy as soon as possible after surgery, within 28 days. Radiotherapy is administered 5 times a week for 6 weeks. Arm II: Within 28 days of surgery, patients receive vincristine IV on days 1, 7, 14, 21, 28, 35, 42, 49, 56, and 63. Carboplatin IV is administered over 1 hour on days 1, 2, 42, and 43. Etoposide IV is administered over 1 hour on days 1-3, 21-23, 42-44, and 63-65. Cyclophosphamide IV is administered over 4 hours on days 21 and 63. As soon as possible after chemotherapy, patients receive radiotherapy as in arm I. Quality of life is assessed every 3 months for the first year and annually thereafter. Patients are followed every 6 weeks for the first year, every 3 months for the second year, every 4 months for the third year, and every 6 months thereafter.

PROJECTED ACCRUAL: A total of 230 patients (115 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven primitive neuroectodermal tumors of the central nervous system No metastatic disease within or outside the central nervous system Must have survived 1 week following surgery Postoperative CT scan and myelogram required

PATIENT CHARACTERISTICS: Age: 3 to 16 Performance status: Not specified Life expectancy: Not specified Hematopoietic: No concurrent hematological disorder Hepatic: Not specified Renal: Renal dysfunction allowed Other: No prior history of malignant disease

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Not specified Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: See Disease Characteristics

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 230 (Estimated)
Dates: Start 1992-04; Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda S. Lashford, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- St. James's Hospital, Leeds, England, United Kingdom

REFERENCES:
- [Result] Taylor RE, Donachie PH, Weston CL, Robinson KJ, Lucraft H, Saran F, Ellison DW, Ironside J, Walker DA, Pizer BL; Children's Cancer and Leukaemia Group CNS Tumour Division. Impact of radiotherapy parameters on outcome for patients with supratentorial primitive neuro-ectodermal tumours entered into the SIOP/UKCCSG PNET 3 study. Radiother Oncol. 2009 Jul;92(1):83-8. doi: 10.1016/j.radonc.2009.02.017. Epub 2009 Mar 26. PMID 19328574
- [Result] Bull KS, Spoudeas HA, Yadegarfar G, Kennedy CR; CCLG. Reduction of health status 7 years after addition of chemotherapy to craniospinal irradiation for medulloblastoma: a follow-up study in PNET 3 trial survivors on behalf of the CCLG (formerly UKCCSG). J Clin Oncol. 2007 Sep 20;25(27):4239-45. doi: 10.1200/JCO.2006.08.7684. PMID 17878477
- [Result] Ellison DW, Onilude OE, Lindsey JC, Lusher ME, Weston CL, Taylor RE, Pearson AD, Clifford SC; United Kingdom Children's Cancer Study Group Brain Tumour Committee. beta-Catenin status predicts a favorable outcome in childhood medulloblastoma: the United Kingdom Children's Cancer Study Group Brain Tumour Committee. J Clin Oncol. 2005 Nov 1;23(31):7951-7. doi: 10.1200/JCO.2005.01.5479. PMID 16258095
- [Result] Lamont JM, McManamy CS, Pearson AD, Clifford SC, Ellison DW. Combined histopathological and molecular cytogenetic stratification of medulloblastoma patients. Clin Cancer Res. 2004 Aug 15;10(16):5482-93. doi: 10.1158/1078-0432.CCR-03-0721. PMID 15328187
- [Result] Taylor RE, Bailey CC, Robinson KJ, Weston CL, Ellison D, Ironside J, Lucraft H, Gilbertson R, Tait DM, Saran F, Walker DA, Pizer BL, Lashford LS; United Kingdom Children's Cancer Study Group Brain Tumour Committee; International Society of Paediatric Oncology. Impact of radiotherapy parameters on outcome in the International Society of Paediatric Oncology/United Kingdom Children's Cancer Study Group PNET-3 study of preradiotherapy chemotherapy for M0-M1 medulloblastoma. Int J Radiat Oncol Biol Phys. 2004 Mar 15;58(4):1184-93. doi: 10.1016/j.ijrobp.2003.08.010. PMID 15001263
- [Result] Taylor RE, Bailey CC, Robinson K, Weston CL, Ellison D, Ironside J, Lucraft H, Gilbertson R, Tait DM, Walker DA, Pizer BL, Imeson J, Lashford LS; International Society of Paediatric Oncology; United Kingdom Children's Cancer Study Group. Results of a randomized study of preradiation chemotherapy versus radiotherapy alone for nonmetastatic medulloblastoma: The International Society of Paediatric Oncology/United Kingdom Children's Cancer Study Group PNET-3 Study. J Clin Oncol. 2003 Apr 15;21(8):1581-91. doi: 10.1200/JCO.2003.05.116. PMID 12697884